CLINICAL TRIAL: NCT00063076
Title: A Two Stage Phase II Randomized Bilateral Comparison of Topical Targretin® Gel 1% in Alopecia Areata
Brief Title: Phase II Randomized Bilateral Comparison of Topical Targretin Gel 1% in Alopecia Areata
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Ligand Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DM02-164
Record Dates: First submitted 2003-06-19; First posted 2003-06-20 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata; Alopecia Totalis; Alopecia Universalis; Targretin Gel
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis | interventions — Bexarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Targretin® (Experimental): Targretin® (bexarotene) Gel 1%, treat half head
  Interventions: Drug: Targretin Gel 1%
- Control (No Intervention): Half head untreated as control

INTERVENTIONS:
Drug: Targretin Gel 1% — Alopecia lesions on one-half of the head including facial hair treated, and other half on head serves as control (untreated). Starting dose once every day till Week 3 then escalate to twice a day.
  Other Names: Targretin
  Arms: Targretin®

SUMMARY:
The goal of this clinical research study is to find the most effective dose of Targretin® (bexarotene) Gel 1% that can be given to patients as a treatment for alopecia areata. The safety and tolerability of this drug will also be studied.

Objectives:

1. Determine the safety and tolerability of Targretin® Gel 1% in the treatment of patients with alopecia areata.
2. Determine the efficacy of Targretin® Gel 1% in the treatment of patients with alopecia areata.

DETAILED DESCRIPTION:
Targretin® (bexarotene) Gel 1% a synthetic vitamin A compound that is approved for the topical treatment and oral treatment of cutaneous T cell lymphoma (CTCL). Vitamin A compounds can influence the growth of skin cells, and can cause the death of T-cells. Researchers hope that the bexarotene may get rid of T-cells around the hair follicles in AA (alopecia areata) lesions.

Before treatment starts, patients will have a complete medical history and a brief physical exam. Researchers will ask about alopecia disease history, date of first diagnosis, and earlier treatments and responses. Blood test (about 4 teaspoons) will be performed before and after the end of treatment. Additional blood tests will be done if needed. Women able to have children must have a negative blood pregnancy test within 7 days before the start of treatment. Blood pregnancy test must be repeated once a month while receiving treatment.

Participants in this study will be randomly assigned (as in the toss of a coin) to treat alopecia areata lesions on only one half of their head. Half of the participants will have the left side treated while the other half will have the right side treated. Sealed envelopes will be given to participants, telling them which side of the head to treat. The other half of the head will remain untreated and serve as the control.

Patients will treat alopecia lesions on one-half of the head including facial hair as designated by the investigator. The other half of the head will have control (untreated) alopecia lesions. Up to 5 index lesions for treatment and 5 control lesions will be designated at baseline to follow and measure during the study. Patients will be treated with Targretin® gel 1% in a dose escalation regimen starting at once every day. At the start of Week 3 patients will begin applications of twice a day applications if tolerated. Patients will continue BID dosing, if tolerated, unless the investigator determines a further increase in application frequency may benefit the patient and the patient agrees to comply.

Patients will be seen at baseline and at weeks 2, 4, 8, 12, 16, 20, 24 and at a 4-week follow-up. Telephone evaluations will be done at week 1 and as needed.

Study visits for evaluation of safety and efficacy will be made at Week 2 and 4 after the start of treatment and then every 4 weeks up until Week 24. Telephone safety evaluations will also be made at Week 1 and other times as needed.

Skin irritation or changes in health during the study may require participants to stop treatment or withdraw from the study.

At withdrawal from the study, about 4 teaspoons of blood will be drawn. The total study duration is 24 Weeks with a 4-week follow-up period. At the 4-week follow-up visit, a physical exam, including measurement of vital signs and weight will be performed. An evaluation of both treated and untreated sides of the head will be performed.

Patients who show a response at 6 months (24 weeks) will be given the option to continue therapy for an additional 6 months and will be able to apply the medication to both sides of the head. Patients will come every 2 months (3 additional visits) and will have the same examination as they have had during the study with evaluation of irritation, hair loss, hair thickness, measurement of lesions, and the physician's global assessment, which is the evaluation of hair re-growth. The same dose adjustment and withdrawal from treatment will be applied during this 6-month period. Every 2 months, blood (about 2 tablespoons) will be drawn for pregnancy tests and to look at your triglycerides (fat) levels and complete blood cell counts.

This is an investigational study. Targretin® Gel 1% is commercially available and approved by the FDA for use in the treatment of cutaneous lesions in patients with CTCL. Initially up to 42 participants will be enrolled in the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of alopecia areata, alopecia totalis, or alopecia universalis.
2. Patients must be 18 years of age to participate.
3. Patients with alopecia areata must have at least two distinct alopecia areata patches >1.0 cm diameter, one located on the right and left sides each of the scalp. Patients with alopecia totalis or universalis will not have distinct alopecia patches but will have complete or total alopecia on both the sides of the scalp. Patients with alopecia totalis or universalis will have one side of the scalp treated. The patient must agree to treat only one side of the scalp with drug, to have photos taken, and to return for follow-up visits.
4. They must also agree to practice two reliable forms of contraception (hormonal, IUD, double barrier) to be used simultaneously unless abstinence is the chosen method during the entire period of treatment and for at least one month after treatment is discontinued.
5. Men with sexual partners who are of childbearing potential or pregnant must use condoms during sexual intercourse during Targretin® gel therapy and for one month after the last application.
6. Patients will be asked to voluntarily contribute pre- and post biopsies for research studies (3 mm punch biopsies for hematoxylin and eosin (H&E) staining and immunohistochemistry of T-cells). However, failure to consent to biopsies will not exclude them from the study.
7. Patients have signed the informed consent.

Exclusion Criteria:

1. Must be off other topical treatment for alopecia areata or PUVA (psoralen + UVA) therapy for at least two weeks.
2. Must have discontinued intralesional steroids or any systemic therapies that are immunosuppressive or that may affect alopecia areata for at least four weeks. Patients who are on chronic oral steroids are not eligible for the study.
3. Women who are pregnant or breastfeeding are excluded. The pregnancy test will be sensitive to at least 25 mlU/ml.
4. Patients with hepatitis, HIV or other serious infections are excluded.
5. Known hypersensitivity to Targretin® drug or to any retinoid or to any ingredient in the study medication.
6. Patients must not have participated in any other investigational drug study within 4 weeks of entry.
7. Patients with Hbg < 9.5 g/dL, WBC < 2,500 K/ul, Platelets < 100 K/ul, TSH > 5.5 or < 0.5 mcU/mL, T4 < 0.9 or > 1.8 g/dl, or fasting triglyceride level > 350 mg/dl will not be eligible to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-05; Primary Completion 2006-10 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Response and toxicity of Targretin Gel 1% treatment for alopecia areata | Baseline and at weeks 2,4,8,12,16,20,24 and at a 4-week follow-up
  "Response" defined as hair growth at PGA grade 3 or 4, and "toxicity" as vesiculation grade 3 or ulceration at grade 4 using design of Thall, Simon and Estey (1995, 1996). To monitor response and toxicity, four possible elementary outcomes are: 1 = [no toxicity, no response], 2 = [no toxicity, response], 3 = [toxicity, no response] , 4 = [toxicity, response].

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Duvic, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org